CLINICAL TRIAL: NCT00156247
Title: Pilot, Single-Arm Study of the Effect of Adding Acitretin to Etanercept Therapy in Patients With Moderate to Severe Psoriasis Who Fail to Respond to Etanercept Monotherapy
Brief Title: Acitretin and Etanercept in Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Collaborators: Connetics Corp. (Unknown)
Responsible Party: Sponsor
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5487
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Results first posted 2015-02-16 (Estimated); Last update posted 2015-02-16 (Estimated); Status verified 2015-02

CONDITIONS: Psoriasis
Keywords: psoriasis; etanercept; acitretin
MeSH Terms: conditions — Psoriasis | interventions — Acitretin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- etanercept with acitretin (Experimental): open-label
  Interventions: Drug: acitretin

INTERVENTIONS:
Drug: acitretin — Patients who have been taking etanercept 50 mg/week for at least 3 months (12 weeks) will take acitretin 25 mg pill once daily for 6 months.
  Other Names: Soriatane

SUMMARY:
To determine whether acitretin plus etanercept is more effective than etanercept alone in clearing psoriasis plaques in adults.

DETAILED DESCRIPTION:
This study will include patients with moderate to severe psoriasis who have been taking etanercept 50 mg/week for at least 3 months (12 weeks) and have not achieved PASI 75. They will be given acitretin 25 mg/day. The combined treatment will occur over 6 months. Subjects' progress will be assessed monthly, based on the improvement of their PASI and PGA scores.

ELIGIBILITY:
Inclusion Criteria:

* Adults (aged 18 to 80 years old) with moderate to severe psoriasis (defined as having a physician global assessment score of 3 [moderate] or higher) who are on etanercept 50 mg SQ once weekly and have not achieved PASI 75 after 12 weeks or more of treatment with etanercept
* All patients on etanercept have been tested for TB before initiation of etanercept

Exclusion Criteria:

* Patients < 18 years old or > 80 years old
* Patients who are not on etanercept 50 mg SQ once weekly
* Women of childbearing potential (Note: women of non-childbearing potential, meaning surgically sterile [bilateral oophorectomy, hysterectomy, and/or bilateral tubal ligation] or post-menopausal for at least 2 years, are eligible)
* Inability to understand consent or comply with study requirements
* Uncontrolled hypertriglyceridemia
* Patients with severely impaired hepatic function
* Patients without health insurance or who are not willing to pay out-of-pocket for etanercept and laboratory tests
* Systemic psoriasis therapies or PUVA within the past 2 weeks
* UVB or topical psoriasis therapies (other than emollients/moisturizers and OTC shampoos) within the past 1 week
* Patients with epilepsy or multiple sclerosis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2005-09; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa A. Magliocco, MD, Principal Investigator — Rutgers, The State University of New Jersey

RESULTS

PARTICIPANT FLOW:
Groups:
- Etanercept With Acitretin: patients on etanercept taking open-label acitretin
Period: Overall Study
Arm/Group | Etanercept With Acitretin
Started | 9
Completed | 5
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Etanercept With Acitretin
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (14.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Percent of Patients Achieving PASI 75 at 6 Months After the Addition of Acitretin Therapy
Description: Percentage of participants achieving at least a 75% decrease (improvement) from Baseline in the Psoriasis Area and Severity Index (PASI) at 6 months. PASI Score incorporates measures of erythema, desquamation, infiltration, and affected body surface area. Involvement and severity of psoriasis was scored using a scale of 0 to 72, where 0 = no psoriasis and 72 = severe disease.
Time Frame: 6 months
Measure: Number; unit: percent
Arm/Group | Etanercept With Acitretin
Number analyzed (Participants) | 8
percent | 12.5

2. Secondary Outcome: Percent of Patients Achieving PASI 50 at 6 Months After the Addition of Acitretin Therapy
Description: Percentage of participants achieving at least a 50% decrease (improvement) from Baseline in the Psoriasis Area and Severity Index (PASI) at 6 months. PASI Score incorporates measures of erythema, desquamation, infiltration, and affected body surface area. Involvement and severity of psoriasis was scored using a scale of 0 to 72, where 0 = no psoriasis and 72 = severe disease.
Time Frame: 6 months
Measure: Number; unit: percent
Arm/Group | Etanercept With Acitretin
Number analyzed (Participants) | 8
percent | 50

3. Secondary Outcome: Percent of Patients Achieving a PGA of Clear or Almost Clear at 6 Months After the Addition of Acitretin Therapy
Description: Percentage of participants achieving a clear (0) or almost clear (1) status on the Physician Global Assessment (PGA) at 6 months. This index evaluates the physician's global assessment of the participant's psoriasis based on severity of induration, scaling, and erythema. The assessment was scored on a scale of 0 to 5, where 0 = clear, with no evidence of plaque elevation, erythema, or scale, and 5 = severe induration, erythema, and scaling.
Time Frame: 6 months
Measure: Number; unit: percent
Arm/Group | Etanercept With Acitretin
Number analyzed (Participants) | 8
percent | 37.5

ADVERSE EVENTS:
Arm/Group | Etanercept With Acitretin
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 2/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Etanercept With Acitretin (N=9)
retinoid dermatitis (Skin and subcutaneous tissue disorders) | 2 (2)
dry/chapped lips (Skin and subcutaneous tissue disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
small sample size; lack of control group

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No